CLINICAL TRIAL: NCT06831643
Title: Standard Volume vs. High Volume Plasma Exchange in Pediatric Acute Liver Failure - A Pilot Randomized Control Trial
Brief Title: Standard Volume vs. High Volume Plasma Exchange in Pediatric Acute Liver Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-ALF-08
Record Dates: First submitted 2025-01-03; First posted 2025-02-18 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Acute Liver Failure
MeSH Terms: conditions — Liver Failure, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SV-TPE group (Experimental): SV-TPE group
  Interventions: Drug: Standard Medical treatment; Biological: Therapeutic Plasma Excahnge
- HV- TPE group (Active Comparator): HV- TPE group
  Interventions: Drug: Standard Medical treatment; Biological: Therapeutic Plasma Excahnge

INTERVENTIONS:
Drug: Standard Medical treatment — Standard Medical treatment
Biological: Therapeutic Plasma Excahnge — Therapeutic Plasma Excahnge

SUMMARY:
Acute liver failure is a multisystem disorder characterized by a syndrome of jaundice, coagulopathy, and encephalopathy with high mortality in the absence of liver transplantation. The pathogenesis of multiorgan failure (MOF) in ALF has been attributed to the release of damage-associated molecular patterns (DAMPs) from injured hepatic cells and microbial pathogen-associated molecular patterns (PAMPs) in the presence of superimposed infection or bacterial translocation.The innate immune cells activated by PAMPs and DAMPs produce pro-inflammatory cytokines [interleukin (IL)-6, IL-1b, IL-8, tumor necrosis factor-alpha (TNF-a)]. Studies indicate that the removal of inflammatory mediators appears to play a role in the treatment of ALF and are removed by some apheresis techniques. Hence therapeutic exchange (TPE) has been used as adjunct or standalone therapy for bridging patients to recovery or LT. TPE to treat liver failure involves two steps-removal of plasma from a patient with liver failure and replacing this with equal volume of fluid; in view of the coagulopathy seen in liver failure patients, the preferred fluid for replacement is fresh frozen plasma. Different doses of PLEX have been used to treat liver failure patients with high, standard or low volume PLEX, to treat ALF. Presently American Apheresis Society guidelines consider High Volume TPE (HV-TPE) as first line the management of ALF. But HV-TPE, apart from strain on blood bank resources (large volumes of fresh frozen plasma needed), also carries risk of transfusion associated acute lung complications, risk of blood borne virus infection, and so on make the use of low-volume PLEX attractive compared to high-volume PLEX. Hence this study is being carried out to consider the safety and efficacy of standard volume plasma exchange (SV-TPE) vs. HV-TPE in Pediatric ALF.

DETAILED DESCRIPTION:
Aim: To study the efficacy in terms of the native liver survival, of standard volume plasma exchange as compared to high volume plasma exchange in Pediatric ALF.

Study Design: Open label pilot Randomized Control trial. Sample size: Time bound. All cases presenting during the study period will be included in the study.

Standard Medical Therapy:

* All patients are were managed by a multidisciplinary team at Live Coma ICU.
* Intubation and ventilation were undertaken for standard indications in addition to the development of grade 3 encephalopathy or evidence of cerebral edema
* Ventilation was managed by fentanyl and propofol along with the use of atracurium for paralysis wherever required.
* Hemodynamics, ONSD and TCD are monitored routinely.
* All patients received N-acetylcysteine.
* Neuro-protective measures such as hypertonic saline, head end elevation, minimal stimulation, propofol and thiopentone infusion are followed as per protocol.
* Anti-ammonia measures like sodium benzoate, CRRT as well started as per protocol.
* CRRT is done for routine renal indications, hyperlactetmia, hyperammonemia.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 3 years to 18 years
2. Fulfilling PALFSG definition (J Pediatr. 2006 May;148(5):652-658).
3. Baseline INR ≥ 2.5, and increasing INR (any value) and/or worsening hepatic. encephalopathy (> 1 grade change) after 6 to 12 hours of standard medical therapy.

Exclusion Criteria:

1. Disseminated intravascular coagulation
2. Marked hemodynamic instability requiring a high dose of vasopressors (norepinephrine >0.5 mcg/kg/min)
3. Signs of irreversible brain injury
4. Any severe cardio-pulmonary pre-existing disease
5. Septic Shock

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Native liver survival at day 21, in patients receiving standard volume (1.3-1.5 times plasma volume) therapeutic plasma exchange and those receiving high volume (2-2.2 times plasma volume) therapeutic plasma exchange in children with acute. | Day 21

SECONDARY OUTCOMES:
Clinical parameters:Grades of Hepatic Encephalopathy from day 0 to day 4. | Day 0,Day1,Day2,day3,Day 4
Clinical parameters: Optic Nerve Sheet Diameter (Left/Right) from day 0 to day 4. | Day 0,Day1,Day2,day3,Day 4
Clinical parameters: Mean arterial pressure from day 0 to day 4. | Day 0,Day1,Day2,day3,Day 4
Proportion of patients with change in Liver Function test from day 0 to day 4. | Day 0,Day1,Day2,day3,Day 4
Biochemical parameters: International normalized ratio from day 0 to day 4. | Day 0,Day1,Day2,day3,Day 4
Biochemical parameters:Arterial ammonia from day 0 to day 4. | Day 0,Day1,Day2,day3,Day 4
Biochemical parameters: Arterial lactate from day 0 to day 4. | Day 0,Day1,Day2,day3,Day 4
Patient with change in Cytokines level at day 0 and day 3. | Day 0 & Day 3
Impact on other factors at day 0 and 3: Growth Factors (G-CSF). | Day 0 & Day 3
Impact on other factors at day 0 and 3: Damage Associated Molecular Pattern (DAMPS) (S100B, HMGB1). | Day 0 & Day 3
Impact on other factors at day 0 and 3: Von Willebrand Factor. | Day 0 & Day 3
Adverse effects in both groups | Within Day 21
Duration of mechanical ventilation & ICU stay. | Within Day 21
Mortality | Within Day 21
Number of participants with Liver Transplant | Within Day 21

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided